CLINICAL TRIAL: NCT01232816
Title: Can T Helper 17 and Regulatory T Cells Explain the Pathophysiology of Delayed Graft Function in Renal Transplant Recipients?
Brief Title: Role of T Helper 17 and Regulatory T Cells in Delayed Graft Function
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Astellas Pharma Canada, Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Steven Paraskevas, Associate Professor of Surgery, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 09-202-SDR
Record Dates: First submitted 2010-10-30; First posted 2010-11-02 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Delayed Graft Function
MeSH Terms: conditions — Delayed Graft Function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine Kidney biopsy Kidney preservation fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Delayed graft function: These are patients in whom dialysis is required following transplantation.
- Immediate function: These are patients in whom no dialysis is required and creatinine declines by >20% in the first 24 hours following transplantation.

SUMMARY:
Delayed graft function (DGF) increases risk of acute rejection after kidney transplantation (KTx). Interleukin-6, which is produced in DGF, is critical in directing naive T helper cells differentiation towards T helper 17 (Th17) and away from regulatory T (Treg) cells. The investigators hypothesize there is an increase in Th17 and a decrease in Treg expression in KTx recipients with DGF compared to those without, leading to immunologic consequences. The investigators will test their hypothesis by measuring in both groups expression of Th17, Treg, and related cytokines in blood, urine, kidney biopsy, and kidney preservation fluid, and correlating these results with immunologic events.

DETAILED DESCRIPTION:
All adult recipients of a primary kidney transplant will be eligible. Subjects will have blood samples drawn from which we will isolate lymphocytes and analyze the Treg population based on surface markers as well as a functional assay. The measures of Treg function will be compared to outcomes including DGF, graft survival and graft function, as well as the development of immunological complications such as donor-specific antibody production, acute rejection, IFTA and opportunistic infection.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipients

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All kidney transplant recipients at our institution will be recruited prior to their operative procedure.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-07; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Graft function | 1 year
  Kidney graft function as measured by GFR

CONTACTS AND LOCATIONS:
Overall Officials: Steven Paraskevas, MD PhD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to make the experimental data available to participants. Their clinical data, however, is available to them through their treating physician.

REFERENCES:
- [Derived] Nguyen MT, Fryml E, Sahakian SK, Liu S, Cantarovich M, Lipman M, Tchervenkov JI, Paraskevas S. Pretransplant Recipient Circulating CD4+CD127lo/- Tumor Necrosis Factor Receptor 2+ Regulatory T Cells: A Surrogate of Regulatory T Cell-Suppressive Function and Predictor of Delayed and Slow Graft Function After Kidney Transplantation. Transplantation. 2016 Feb;100(2):314-24. doi: 10.1097/TP.0000000000000942. PMID 26425877